CLINICAL TRIAL: NCT06024551
Title: Investigation of the Efficacy of Telerehabilitation in Patients With Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Associate Professor, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TR35TR
Record Dates: First submitted 2023-04-04; First posted 2023-09-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Injuries; Rotator Cuff Tendinitis
Keywords: rotator cuff tendinopathy; telerehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients who receive telerehabilitation
  Interventions: Other: Telerehabilitation
- Control Group (Other): Patients who receive home exercise program
  Interventions: Other: home exercise program

INTERVENTIONS:
Other: Telerehabilitation — Patients in this arm will be given telerehabilitation three times a week, for four weeks.
  Arms: Intervention Group
Other: home exercise program — Patients in this arm will receive home exercise program for four weeks
  Arms: Control Group

SUMMARY:
The goal of this study is to investigate the effect of telerehabilitation in patients with rotator cuff tendinopathy. The main questions it aims to answer are:

* Is telerehabilitation effective in improving the functional status of patients with rotator cuff tendinopathy?
* Is telerehabilitation effective in reducing the pain of rotator cuff patients?

DETAILED DESCRIPTION:
Patients between the ages of 18-65 who were diagnosed with rotator cuff tendinopathy will be included in the study. Patients will be divided into two groups. Patients in group 1 will be given a home exercise program. Then, the patients will be called 3 times a week and it will be evaluated whether they do their exercises regularly and whether they do it correctly. At the end of the first month, the patients will be evaluated again for functionality and pain.

The patients in group 2 will be given a home exercise program and at the end of the first month, the patients will be evaluated again in terms of functionality and pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rotator cuff tendinopathy
* Being able to do the prescribed exercises
* Having an access to internet and having a computer or smart phone for telerehabilitation

Exclusion Criteria:

* Patients with a neurological disease that may affect the effectiveness of exercise
* History of fracture in shoulder region
* History of surgery in shoulder region
* Patients with a psychiatric disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index | one month
  Western Ontario Rotator Cuff Index is a disease-specific quality of life questionnaire, evaluating the change in symptoms and functional ability, specific to a Rotator Cuff tendinopathy. Raw scores range from 0 to 2100 with a higher score indicating decreased quality of life.
Simple Shoulder Test | one month
  A questionnaire about the function of the involved shoulder. Overall scored is calculated by number of yes/number of completed items. Minimum score is 0 %and maximum is 100 %. Higher scores indicate better function.

SECONDARY OUTCOMES:
Range of motion | one month
  Shoulder joint normal range of motion will be measured using a goniometer. Normal movements of the shoulder joint are flexion 180 degrees, abduction 180 degrees, hyperextension 45 degrees, internal rotation 70 degrees and external rotation 90 degrees. Limitations will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ferruh Taşpınar, Study Director — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)